CLINICAL TRIAL: NCT05434377
Title: A Randomized Study Comparing Between Fixed Dose and Serum Level-Based Titration Regimen of Vitamin D Supplementation Among Dialysis Patients
Brief Title: A Study of Fixed Dose Versus Serum Level-Based Titration Regimen of Vitamin D Supplementation in Dialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Piyawan Kittiskulnam, Associate Professor of Medicine, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 326/65
Record Dates: First submitted 2022-06-21; First posted 2022-06-28 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Vitamin D Deficiency; End Stage Renal Disease
Keywords: vitamin D insufficiency; dialysis; ergocalciferol
MeSH Terms: conditions — Vitamin D Deficiency; Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D supplementation using titration regimen (Active Comparator): Patients will receive ergocalciferol orally depending on serum 25(OH)D level as described
  * serum 25(OH)D < 5 ng/ml --> receive ergocalciferol 50,000 IU/week for 3 months followed by 50,000 IU monthly for 3 months
  * serum 25(OH)D 5-15 ng/ml--> receive ergocalciferol 50,000 IU/week for 1 month followed by 50,000 IU monthly for 5 months
  * serum 25(OH)D 16-30 ng/ml--> receive ergocalciferol 50,000 IU monthly for 6 months
  Interventions: Other: ergocalciferol supplementation; Other: dialysis techniques; Other: sunlight exposure time
- Vitamin D supplementation using fixed dose regimen (Experimental): Patients will receive ergocalciferol 20,000 unit orally per week for 6 months.
  Interventions: Other: ergocalciferol supplementation; Other: dialysis techniques; Other: sunlight exposure time

INTERVENTIONS:
Other: ergocalciferol supplementation — Participants in both groups will recieve ergocalciferol with different supplementation regimens for 6 months.
  Other Names: nutritional vitamin D supplementation
Other: dialysis techniques — Both groups will have participants treated with maintenance hemodialysis and peritoneal dialysis.
  Other Names: mode of dialysis
Other: sunlight exposure time — Both groups will be advised to receive similar hours of daily sunlight exposure time.

SUMMARY:
Vitamin D insufficiency, defined as serum 25-hydroxyvitamin (OH) D level less than 30 ng/ml, is highly prevalent not only in the general population but also in chronic kidney disease (CKD) population. Many guidelines including the National Kidney Foundation-Kidney Disease Outcomes Quality Initiative (NKF-KDOQI) have consistently recommended vitamin D supplementation in patients with pre-dialysis CKD with vitamin D insufficiency with ergocalciferol or cholecalciferol to achieve 25(OH)D level of more than 30 ng/ml using serum levels-based titration regimen. However, this protocol has not been studied in end stage kidney disease patients treated with maintenance dialysis.

DETAILED DESCRIPTION:
The investigators plan to conduct a randomized study comparing the two different protocols between serum 25(OH)D level-based titration regimen and fixed dose of ergocalciferol supplementation among dialysis patients for a total period of 6 months. At the study completion, investigators also plan to compare the proportion of participants achieving serum 25(OH)D of more than 30 ng/ml, CKD-related metabolic and bone parameters as well as non-skeletal effect of vitamin D supplementation for each group.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* on maintenance dialysis (hemodialysis or peritoneal dialysis) > 3 months
* 25(OH)D < 30 ng/ml
* able to provide inform consent form

Exclusion Criteria:

* current ergocalciferol or cholecalciferol treatment
* known allergy to ergocalciferol
* active inflammation or infection
* advanced stage of cancer
* pregnancy
* lactation
* on immunosuppressive drugs or corticosteroids

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
proportion of patients with vitamin D adequacy | 6 months
  serum 25(OH)D more than 30 ng/ml

SECONDARY OUTCOMES:
serum calcium | 6 months
  pre-dialysis serum calcium levels
serum phosphorus | 6 months
  pre-dialysis serum phosphorus levels
serum intact parathyroid hormone | 6 months
  pre-dialysis serum intact parathyroid hormone levels
muscle mass | 6 months
  bioimpedance-derived muscle mass measurement
muscle strength | 6 months
  handgrip strength measurement

CONTACTS AND LOCATIONS:
Overall Officials: Piyawan Kittiskulnam, Principal Investigator — Chulalongkorn University
Locations (1):
- Chulalongkorn Univeristy, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No